CLINICAL TRIAL: NCT06362967
Title: The Efficacy and Safety of Immunosorbent or Plasma Exchange Combined With Rituximab and High-dose IVIG for Patients With High Titers of Anti-HLA Antibodies Prior to Allogeneic Hematopoietic Stem Cell Transplantation: A Single-Centre, Single-Arm, Phase II Clinical Study
Brief Title: The Efficacy and Safety of Desensitation Regimen for Patients With High Titers of Anti-HLA Antibodies Prior to Allo-HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-HLA antibody
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: High Titers of Anti-HLA Antibody (MFI ≥5000)
Keywords: immunoadsorption or plasma exchange；rituximab；high-dose IVIG
MeSH Terms: interventions — Rituximab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- antibody desensitisation group (Experimental): Immunoadsorption or plasma exchange combined with rituximab, high-dose IVIG
  Interventions: Combination Product: Immunoadsorption or plasma exchange combined with rituximab, high-dose IVIG

INTERVENTIONS:
Combination Product: Immunoadsorption or plasma exchange combined with rituximab, high-dose IVIG — For allogeneic haematopoietic stem cell transplantation patients with high titers of anti-HLA antibodies present in the body, a desensitisation regimen of immunosorbent or plasma exchange combined with rituximab and high-dose IVIG is used prior to transplantation.
  Other Names: Intravenous Immunoglobin

SUMMARY:
Evaluation of the efficacy and safety of immunoadsorption or plasma exchange combined with rituximab and high-dose IVIG to reduce high titres of anti-HLA antibodies in patients prior to allogeneic haematopoietic stem cell transplantation

DETAILED DESCRIPTION:
Approximately 10-21% of allogeneic hematopoietic stem cell transplantation (allo-HSCT) patients have non-specific or donor-specific anti-HLA antibodies (DSAs) prior to transplantation. Patients with combined DSAs and mean fluorescence intensity (MFI) ≥ 5000 can lead to a significantly higher incidence of primary graft failure and graft dysfunction after transplantation, and increased transplant-related mortality (TRM). Meanwhile, a retrospective study at our centre found that patients with high titre non-specific antibodies (MFI ≥ 5000) present before cord blood transplantation had significantly higher TRM in the early post-transplantation period. Therefore, our centre intends to conduct a single-arm prospective cohort study to explore whether the desensitisation regimen of immunosorbent or plasma exchange combined with rituximab and high-dose IVIG before transplantation in allogeneic hematopoietic stem cell transplantation patients with high titres of anti-HLA antibodies can lower the antibody titres in the patient's body, reduce the incidence of transplant-related complications, and improve the prognosis of transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects to undergo allo-HSCT
2. Age 14-60, No gender, No ethnicity
3. ECOG score ≤ 2
4. Population reactive antibody screening within 1 month prior to transplantation HLA-class I or class II antibody MFI ≥ 5000
5. No severe organ failure and no active infections
6. Subjects and their families voluntarily undergo anti-HLA antibody testing and antibody desensitisation treatment and sign an informed consent form

Exclusion Criteria:

1. Those with severe organ dysfunction or disease, such as severe disease and dysfunction of the heart, liver, kidneys and pancreas
2. Pregnancy
3. Subjects and/or authorised family members who refuse to accept antibody desensitisation treatment
4. Persons with any life-threatening disease, physical condition, or organ system dysfunction that, in the opinion of the investigator, may compromise the safety of the subject and place the results of the study at unnecessary risk
5. Persons with drug dependence,uncontrolled psychiatric disorders and persons with cognitive dysfunction
6. Participants in other clinical studies within 3 months
7. Those whom the investigator considers unsuitable for enrolment (e.g., subjects will not be able to adhere to examinations and treatments due to financial or other issues)

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of reduction of anti-HLA antibody MFI values to less than 5000 in subjects at the end of treatment | at the end of desensitation treatment
  Incidence of reduction of anti-HLA antibody MFI values to less than 5000 in subjects at the end of treatment

SECONDARY OUTCOMES:
Incidence of primary graft failure | 42 days
  Incidence of primary graft failure
Incidence of TRM after allo-HSCT | 100 days
  Incidence of TRM after allo-HSCT
Incidence of ineffective platelet transfusion after allo-HSCT | 100 days
  Incidence of ineffective platelet transfusion after allo-HSCT
Cumulative incidence of neutrophil engraftment after allo-HSCT | 42 dyas
  Cumulative incidence of neutrophil engraftment after allo-HSCT cumulative incidence of neutrophil engraftment after allo-HSCT
Cumulative incidence of II-IV° acute GVHD | 100 days
  Cumulative incidence of II-IV° acute GVHD
Cumulative incidence of relapse at 1 year post-transplant | 360 days
  Cumulative incidence of relapse at 1 year post-transplant
Probability of overall survival post transplantation | 360 days
  Probability of overall survival post transplantation
Incidence of allergies and allergic reactions | at the end of desensitation treatment
  Incidence of allergies and allergic reactions
Incidence of haemorrhagic events | at the end of desensitation treatment
  Incidence of haemorrhagic events
Incidence of viral, bacterial and fungal infections | at the end of desensitation treatment
  Incidence of viral, bacterial and fungal infections
Incidence of hypocalcaemia | at the end of desensitation treatment
  Incidence of hypocalcaemia

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, ph.D., Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No